CLINICAL TRIAL: NCT02267200
Title: The Screening and Analysis of Plasma Biomarkers in Irreversible Pulmonary Arterial Hypertension Associated With Congenital Heart Disease
Brief Title: The Screening and Analysis of Plasma Biomarkers in Irreversible PAH-CHD
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhuoming, Vice Chief, Department of thoracic and cardiovascular surgery, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SCMCIRB-K2014004
Record Dates: First submitted 2014-09-25; First posted 2014-10-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension,Pulmonary
Keywords: biomarkers，pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- reversible PAH group: reversible PAH was defined as sPAP decreasing to 40 mmHg after follow-up more than 6 months through echocardiography.
- irreversible PAH group: irreversible PAH was defined as 6 months after surgery through echocardiography ，the sPAP remaining 40 mmHg or up

SUMMARY:
The purpose of this study is to analyse the sensitivity and specificity of circulating endothelial cells to predict irreversible pulmonary arterial hypertension associated with congenital heart disease.

DETAILED DESCRIPTION:
predict to recruit 100 patients with pulmonary arterial hypertension (PAH)associated with CHD，under the commitment of the children's parents，take 3-4ml central venous blood before the corrective surgery，then calculate the number of the circulating endothelial cells by flow cytometer AND detect the expression of micro RNAs to screen out the biomarker，through the 6 months follow-up, separated the reversible and irreversible PAH,then to carry on the statistics.

ELIGIBILITY:
Inclusion Criteria:

* Only those patients with systolic PAP (sPAP) >65mmHg before surgery were included.

Exclusion Criteria:

* Patients with trisomy 21 (Down syndrome) were not included

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: those patients with systolic PAP (sPAP) >65mmHg before surgery were included.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
the number of Circulation endothelial cells and the detective count of microRNAs | 6 months after corrective surgery
  the number of Circulation endothelial cells and the detective count of microRNAs in the biomarkers in both groups differd significantly.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoming Xu, Ph D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China